CLINICAL TRIAL: NCT02403232
Title: Autologous Adipose-derived Stem Cells (ASCs) for the Treatment of Perianal Fistula in Crohn Disease: A Pilot Study
Acronym: ASPEFIC1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bertoli, MD, Papa Giovanni XXIII Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Perianal Fistula; Crohn Disease
Keywords: Autologous adipose-derived stem cells
MeSH Terms: conditions — Crohn Disease

ARMS (1):
- ASCs injection (Experimental): Autologous adipose-derived stem cells (ASCs) injection with LIPOGEMS system.
  Interventions: Procedure: ASCs injection; Device: ASCs injection; Device: Closure of fistula tract.

INTERVENTIONS:
Procedure: ASCs injection — In the infiltration step, adrenalin in a saline solution is infiltrated using a 19-cm specially designed disposable blunt cannula.
  The aspiration step is performed by a luer-lock syringe connected to a disposable 19-cm blunt cannula.
  The harvested lipoaspirate can be progressively put into the device using multiple 10-cc syringes.
  Subsequently, in lithotomy position, a seton will be removed and a fistula tract will be thoroughly curetted and irrigated. After a mucosal flap preparing round the internal opening, cells will be injected in the perianal adipose tissue.
Device: ASCs injection — In general anesthesia subcutaneous abdominal adipose tissue will be collected by LIPOGEMS system to prepare ASCS.
  Other Names: LIPOGEMS system
Device: Closure of fistula tract. — A SALVECOLL-E paste will be injected into the fistula tract.
  Other Names: SALVECOLL-E paste

SUMMARY:
Crohn's disease is an immunologically mediated inflammatory bowel disease with a reported incidence of 4.0-7.0, 7.1, and 1.34 per 100,000 persons in Europe, the U.S., and Korea, respectively. Uncontrolled chronic inflammation finally causes various complications in intestine such as bowel obstruction, fistulas, abscesses, and anal fissures.

The incidence of perianal fistula was reported in 13%- 39% of patients with Crohn's disease. Medical treatment for Crohn's fistulae initially focused on surgical intervention accompanied by symptomatic treatment with antibiotics and immunosuppressants. The most serious problem after surgical intervention is the relatively high incidence of postoperative anal incontinence caused by sphincter injury during the procedure. Conversely, available pharmacological therapies for Crohn's fistulae based on biologic agents such as infliximab do not generally reach ideal goal of treatment (e.g., complete closure of the fistula). A high recurrence rate after treatment with infliximab has also been reported, even after long-term maintenance therapy, which suggests that infliximab monotherapy does not provide adequate healing.

The ACCENT II study demonstraded a complete fistula healing in 25% of patients. To reach a better clinical outcome, combination treatment with infliximab and surgical intervention is highly recommended for management of Crohn's fistulae. Nonetheless, even this strategy does not result in a satisfactory healing for many patients.

The ideal therapeutic goal of treatment is not only complete closure of the fistula without recurrence but also preservation of anal sphincter function. Unfortunately, currently available medical or surgical treatment is not likely to offer a cure for perianal fistulae and, as noted above, recurrence is frequently reported.

Together with active research in the field of bone marrow-derived mesenchymal stem cells (BM-MSCs) and hematopoietic stem cells, autologous or allogenic adipose tissue-derived stem cells (ASCs) have been studied for management of Crohn's disease and other disorders.

Of particular relevance to this study, ASCs could be considered to be safe and efficacious therapeutic tools for the treatment of Crohn's fistulae. Importantly, ASCs do not cause fecal incontinence after injection into the lesion site in Crohn's disease patients. A phase I dose-escalation clinical study with ASCs manufactured by Anterogen Co., Ltd. (Seoul, Korea) demonstrated the safety and therapeutic potential of these cells for the treatment of Crohn's fistulae. A phase II study demonstrated a good rate of cronh's related fistula closure using a ASCS injection.

Actually the best accepted treatment of Crohn related perianal fistula, is the surgical procedure in association whit medical therapy.

DETAILED DESCRIPTION:
Basic information:

Lipogems: Lipogems® system is a disposable device for liposuction, processing and adipose tissue reinjection. Procedure takes place in a single surgical time. It's a disposable device that progressively reduces adipose tissue clusters size, washing completely pro-inflammatory oil and blood debrides through a minimal manipulation "free enzyme" in a aseptic closed system completely preﬁlled by room temperature physiological solution.

Lipogems product is a non-expanded and microfractured fat tissue ready for autologous settings.

SalveColl-E: Salvecoll® is sterile bioplastic, equine derived, type I collagen material with a fully preserved fibrous structure (non-reconstructed) that ensures the regeneration of affected tissues. Type I collagen has zero risk of transmitting viral or microbial infections.

Rationale for the trial: To evaluate the efficacy of the use of ACSS in crohn related perianal fistulas. The aim of the study is to improve fistula healing at 1 year from 25% to 65%.

Treatment of subjects At the time of fistula diagnosis the patients will be screened for eligibility and a informed consent will be administered . All patients will be underwent a loose seton placement after antibiotics prophylaxis administration with Ciprofloxacin and Metronidazole to obtain a pelvis sepsis resolution at time 0.

At week 4 a surgical procedure will be performed. In general anesthesia a antibiotics prophylaxis will be administrated and subcutaneous abdominal adipose tissue will be collected by LIPOGEMS system to prepare ASCS.

In the infiltration step, adrenalin in a saline solution (2 μg/ml final concentration) is infiltrated using a 19-cm specially designed disposable blunt cannula.

The vasoconstriction together with the blunt point of the cannula avoids any accidental intravascular injection and facilitates the subsequent lipoaspiration. Three hundred to 500 ml are usually injected in the chosen area for fat harvesting (usually the lower abdomen), making the tissue really "filled" with the injecting solution. The aspiration step (lipoaspirate) is performed by a luer lock syringe connected to a disposable 19-cm blunt cannula (3 mm OD), with 5 oval holes (1 ´ 2 mm). A few strokes using a standard liposuction technique are enough to harvest 6-10 ml of fat tissue. Vacuum while aspirating can be obtained manually or by clamping the syringe plunger with a clamp instrument. Up to 1,000 ml can be harvested in less than 15 min, and 1-2 min are enough. The harvested lipoaspirate can be progressively put into the device using multiple 10-cc syringes.

Subsequently, in lithotomy position, a seton will be removed and a fistula tract will be thoroughly curetted and irrigated. After a mucosal flap preparing round the internal opening, cells will be injected in the perianal adipose tissue.

Between 40 and 130 ml of lipoaspirate (ideally 100 ml) are processed at each time in the standard 225-ml device. To avoid cell damage, no air should be in the device during all procedural steps and the device should be prefilled with saline before beginning the processing. The aspirated fat should be always surrounded by a liquid environment: this is essential to obtain healthy smaller fat clusters instead of oil and adipose tissue debris. The first cluster reduction was obtained by pushing the aspirated fat from the syringe into the device and through the first size reduction filter while allowing the corresponding quantity of saline to exit towards the waste bag. The final Lipogems product is then collected into 10-ml syringes connected to the upper opening of the device. The final Lipogems product is now ready for the injection in the perianal fistula.

After a SALVECOLL-E paste injection into the fistula tract the mucosal flap will may be closed with an absorbable interrupted sutures. A external opening will be sealed with Dermabond Mini.

The patients will receive a intravenous infusion of Infliximab (Remicade) at a dose of 5 mg per kilogram of body weight at weeks 8, 10, 14 and every 8 week for a total of nine doses.

Rationale for treatment The ASCS injection in the perianal adipose tissue in association with Infliximab therapy, would improve a crohn related perianal fistula healing.

This association could be reduce a recurrence and reintervention rate with an improvement of quality of life.

Trial population Number of subjects to be studied Planned number of subjects to be screened: 10 Anticipated number of trial sites: 1

Withdrawal criteria The subject may withdraw at will at any time. The patient may be withdrawn from the trial at the discretion of the investigator for safety concerns. If the patient withdraws or is withdrawn at any time after receiving trial product, final safety information will be obtained.

Patients who are deemed during surgery not suitable included in this protocol will be withdrawn from the study. In case a subject is being prematurely withdrawn from the trial the Investigator will ensure that the procedures for the last visit are undertaken, if possible. The primary reason (adverse event, non-compliance with protocol or other) for discontinuation must be specified in the CRF.

A patient withdrawn from the study will be analyzed according to evaluability of Subjects for Analysis.

Methods and assessments Visit procedures

The study comprises of the following visits:

* Visit 1: Diagnosis, baseline visit and first surgery procedure: Screening of patient, Baseline examination, Pre-surgery and surgery assessment, Informed consent.
* Visit 2: Treatment visit: Surgery
* Visit 3: Medical treatment: start Infliximab administration
* Visit 4, 5, 6, 7,8,9: Medical treatment follow-up
* Visit 10: end of study: last infliximab dose

In case of any premature discontinuation of the trial, the patient will, if possible, be called in for a last visit. Even if the patient is not able to attend, the End of Trial Form must be completed.

The Investigator must keep a subject screening log and a subject enrolment log. These can be combined in one document.

Subjects enrolled in the trial will be provided with a documents stating that he/she is in a trial, contact address and telephone numbers.

In case a subject is being prematurely withdrawn from the trial the Investigator will ensure that the procedures for the last visit are undertaken, if possible. The primary reason (adverse event, non-compliance with protocol or other) for discontinuation must be specified in the CRF.

All patients will be classified according to the American Society of Anesthesiology Physical Status Classification as described below. No restriction regarding to ASA status will be applied in this trial.

Patient Compliance The investigator will reinforce compliance with the protocol by ensuring that only patients willing to follow the trial procedures are enrolled in the trial.

Definitions adverse events

Adverse event (AE):

Any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.

An adverse event can therefore be any unfavourable and unintended sign (e.g., including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Note: This includes events from the first trial related activity after the subject has signed the informed consent and until post treatment follow-up period as defined in the protocol.

The following should not be recorded as AEs:

* Pre-planned procedures unless the condition for which the procedure was planned has worsened from the first trial related activity after the subject has signed the informed consent.
* Pre-existing conditions found as a result of screening procedures. These should be recorded as medical history/concomitant illness.

An AE can also be a clinical laboratory abnormality regarded as clinically significant i.e. an abnormality that suggests a disease and/or organ toxicity and is of a severity which requires active management (i.e. discontinuation of trial product, more frequent follow-up or diagnostic investigation).

The following events will not be recorded as adverse events, as such discomforts are expected to be related to the surgical procedure:

* Post operative nausea/vomit
* Post operative sore throat due to intubation
* Post operative pain due to surgical intervention within 3 months from the operation.

Serious adverse event (SAE):

A SAE is an experience that at any dose results in any of the following:

* Death
* A life-threatening* experience
* In-subject hospitalization or prolongation of existing hospitalization
* A persistent or significant disability/incapacity
* Important medical events that may not result in death, be life-threatening*, or require hospitalization may be considered a SAE when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

  * The term "life-threatening" in the definition of SAE refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event which hypothetically might have caused death if it was more severe.

Non-serious adverse event:

A non-serious AE is any AE which does not fulfil the definition of a serious AE.

Severity assessment definitions:

* Mild - No or transient symptoms, no interference with the subject's daily activities.
* Moderate - Marked symptoms, moderate interference with the subject's daily activities.
* Severe - Considerable interference with the subject's daily activities, unacceptable.

Relationship to trial product assessment definitions:

* Probable: good reasons and sufficient documentation to assume a causal relationship
* Possible: a causal relationship is conceivable and cannot be dismissed
* Unlikely: the event is most likely related to an aetiology other than the trial product

Outcome categories and definitions:

* Recovered - Fully recovered, or by medical or surgical treatment the condition has returned to the level observed at the first trial related activity after the subject signed the informed consent.
* Recovering - The condition is improving and the subject is expected to recover from the event. This term should only be used when the subject has completed the trial.
* Recovered with sequelae - As a result of the AE the subject suffered persistent and significant disability/incapacity (e.g. became blind, deaf, paralyzed). Any AE recovered with sequelae should be rated as an SAE.
* Not recovered.
* Fatal.
* Unknown - This term should only be used in cases where the subject i

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years old
* Diagnosis of perianal fistulae associated with Crohn's disease.

Exclusion Criteria:

* Patients aged < 18 years old
* Informed consent refusal
* Medical or family history of variant Creutzfeldt-Jakobs disease
* Activated sever Crohn's disease
* Perianal fistulae >2 cm in diameter
* Autoimmune disease or inflammatory bowel disease other than Crohn's disease
* Infectious disease including hepatitis B virus, hepatitis C virus and immunodeficiency virus infection
* Active tuberculosis
* Signs of septicemia
* Patients treated with Infliximab within 3 months prior to ASC treatment.
* Technically difficult adipose tissue collection due to low levels of fat tissue.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Healing fistula | 62 weeks

SECONDARY OUTCOMES:
Morbidity | 62 week
Quality of life modification | 62 week
Relation between Crohns Disease Activity Index and fistula healing | 62 week
Mortality | 62 week

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Bertoli, Bergamo, Italy, Italy